CLINICAL TRIAL: NCT03743025
Title: Metabolic Phenotyping During Stress Hyperglycemia in Cardiac Surgery Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was terminated following the Data and Safety Monitoring Board (DSMB) review due to concerns with perioperative use of the study drug.
Sponsor: Emory University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Francisco Pasquel, Associate Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00097963; 1K23GM128221-01A1 (NIH)
Record Dates: First submitted 2018-11-14; First posted 2018-11-15 (Actual); Results first posted 2024-05-30 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Stress Hyperglycemia
Keywords: Coronary Artery Bypass Surgery (CABG); Post Operative; Obesity
MeSH Terms: conditions — Obesity | interventions — dulaglutide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: Prospective placebo controlled randomized study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Dulaglutide Arm (Experimental): Participants without a history of DM who are randomized to receive a single injection of dulaglutide (0.75 mg/0.5 mL solution in a single-dose pen) one to three days prior to surgery.
  Interventions: Drug: Dulaglutide Injection
- Placebo Arm (Placebo Comparator): Participants without a history of DM who are randomized to receive a single injection of a placebo (saline injection of 0.5 mL pre-drawn solution) one to three days prior to surgery.
  Interventions: Other: Saline Injection

INTERVENTIONS:
Drug: Dulaglutide Injection — Participants randomized at pre-surgery/anesthesia visit and without a history of DM will receive a single injection of Dulaglutide injection: 0.75 mg/0.5 mL solution in a single-dose pen 1 to 3 days prior to surgery
  Other Names: Trulicity
  Arms: Dulaglutide Arm
Other: Saline Injection — Participants randomized at pre-surgery/anesthesia visit and without a history of DM will receive a single injection of Saline injection/0.5 mL pre-drawn solution 1 to 3 days prior to surgery
  Other Names: Sodium Chloride Injection
  Arms: Placebo Arm

SUMMARY:
This study is a prospective randomized study to examine the effects of exposure to dulaglutide on the prevention of stress-hyperglycemia and the metabolic inflammatory response in the perioperative period.

DETAILED DESCRIPTION:
Stress hyperglycemia is common in the perioperative period and is associated with increased risk of death postoperatively. Counterregulatory hormones and inflammatory mediators appear to modulate the acute biological response to stress, however, the pathophysiological pathways that result in stress hyperglycemia and its link to poor clinical outcomes are not well understood. At least half of non-diabetes mellitus (DM) patients undergoing cardiac surgery develop stress hyperglycemia shown to be an independent risk factor of morbidity and mortality. The current approach to treat hyperglycemia with insulin has major limitations including high resource utilization and high risk of hypoglycemia. The main goals of this study are to examine baseline and postoperative metabolic profiles of non-diabetic, coronary artery bypass grafting (CABG) patients with stress hyperglycemia and to study the effect of a long-acting glucagon-like peptide-1 receptor agonists (GLP-1 RA) on the prevention of stress-hyperglycemia and modulation of metabolic stress during cardiac surgery.

To examine whether exposure to dulaglutide, a GLP-1 RA, can improve glycemic control and ameliorate the inflammatory response to acute surgical stress, obese patients without diabetes mellitus undergoing CABG surgery will be randomized to receive either dulaglutide or placebo two to three days prior to surgery. The researchers of this study ultimately want to provide evidence to support the use of novel therapies to prevent and manage stress hyperglycemia in the inpatient setting.

ELIGIBILITY:
Inclusion Criteria:

* Males or females between the ages of 40 and 80 years
* Body mass index (BMI) ≥25
* Undergoing elective CABG surgery
* No previous history of diabetes or hyperglycemia

Exclusion Criteria:

* Hyperglycemia (BG>125 mg/dl or HbA1c > 6.5%) or previous treatment with antidiabetic agents
* Impaired renal function (GFR < 30 ml/min) or clinically significant hepatic failure
* Gastrointestinal obstruction expected to require gastrointestinal suction
* Patients with clinically relevant pancreatic or gallbladder disease
* Treatment with oral or injectable corticosteroid
* Mental condition rendering the subject unable to understand the possible consequences of the study
* Pregnancy or breastfeeding at time of enrollment

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-03-08 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Pasquel, MD, MPH, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Emory Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from Grady Memorial Hospital, Emory University Hospital Midtown, and Emory University Hospital in Atlanta, Georgia, USA. Participant enrollment began March 8, 2019 and the final study assessment occurred on May 2, 2023.
Groups:
- Dulaglutide: Participants without a history of diabetes mellitus (DM) who were randomized to receive a single injection of dulaglutide (0.75 mg/0.5 mL solution in a single-dose pen) one to three days prior to elective coronary artery bypass graft (CABG) surgery.
- Placebo: Participants without a history of DM who were randomized to receive a single injection of a placebo (saline injection of 0.5 mL pre-drawn solution) one to three days prior to elective CABG surgery.
Period: Overall Study
Arm/Group | Dulaglutide | Placebo
Started | 14 | 14
Completed | 12 | 13
Not Completed | 2 | 1
Not completed — Surgery was cancelled | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Dulaglutide: Participants without a history of DM who were randomized to receive a single injection of dulaglutide (0.75 mg/0.5 mL solution in a single-dose pen) one to three days prior to surgery.
- Placebo: Participants without a history of DM who were randomized to receive a single injection of a placebo (saline injection of 0.5 mL pre-drawn solution) one to three days prior to surgery.
- Total: Total of all reporting groups
Arm/Group | Dulaglutide | Placebo | Total
Number analyzed (Participants) | 14 | 14 | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 8 | 19
  >=65 years | 3 | 6 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.00 (11.62) | 61.50 (10.86) | 59.40 (10.87)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 1 | 4
  Male | 11 | 13 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 14 | 12 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 2 | 5
  White | 11 | 12 | 23
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14 | 14 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Blood Glucose Levels (BG) > 140 mg/dl During Post Operative Period
Description: Stress-hyperglycemia is defined as any post-CABG hospital-obtained blood glucose (BG) levels >140 milligrams per deciliter (mg/dL). Information on BG measurements was collected both at bedside by glucose meter and by hospital laboratory. BG was measured every 1-2 hours during continuous insulin infusion (CII) in the ICU, and before meals and at bedtime after transition to regular wards.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
Participants | 11 | 13

2. Secondary Outcome: Mean Blood Glucose Levels During the Intensive Care Unit (ICU) Stay Postoperatively
Description: To measure glucose control, the mean blood glucose levels in mg/dL were measured during the postoperative Intensive Care Unit (ICU) stay. Information on BG measurements was collected both at bedside by glucose meter and by hospital laboratory. BG was measured every 1-2 hours during continuous insulin infusion (CII) in the ICU, and before meals and at bedtime after transition to regular wards.
Time Frame: During the ICU stay (up to 7 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
mg/dL | 134.11 (14.00) | 129.79 (11.42)

3. Secondary Outcome: Number of Participants Needing CII Treatment in the ICU
Description: Patients with two consecutive BG >180 mg/dl, or average daily BG >180 mg/dl were started on rescue therapy with subcutaneous basal insulin (glargine or levemir) once daily. Information on BG measurements was collected both at bedside by glucose meter and by hospital laboratory. BG was measured every 1-2 hours during continuous insulin infusion (CII) in the ICU, and before meals and at bedtime after transition to regular wards. The number of participants needing CII while in the ICU postoperatively was compared between patients randomized to dulaglutide or placebo study arms.
Time Frame: During the ICU stay (up to 7 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
Participants | 11 | 12

4. Secondary Outcome: Number of Participants With Stress-hyperglycemia Requiring Rescue Therapy With Subcutaneous Insulin After Discontinuation of CII
Description: Patients with two consecutive BG >180 mg/dl, or an average daily BG >180 mg/dl were started on rescue therapy with subcutaneous basal insulin (glargine or levemir) once daily. Information on BG measurements was collected both at bedside by glucose meter and by hospital laboratory. BG was measured every 1-2 hours during continuous insulin infusion (CII) in the ICU, and before meals and at bedtime after transition to regular wards. The number of participants in need of rescue therapy with subcutaneous insulin postoperatively, after CII was discontinued, was compared between study arms.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who required CII while in the ICU.
Measure: Count of Participants; unit: Participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 11 | 12
Participants | 6 | 4

5. Secondary Outcome: Mean Blood Glucose Levels During the Hospital Stay
Description: To measure glucose control, the mean blood glucose levels in mg/dL during the non-ICU hospital stay postoperatively were measured. Information on BG measurements was collected both at bedside by glucose meter and by hospital laboratory. BG was measured every 1-2 hours during continuous insulin infusion (CII) in the ICU, and before meals and at bedtime after transition to regular wards.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
mg/dL | 119.69 (23.50) | 117.69 (20.59)

6. Secondary Outcome: Mean Units Per Hour of Insulin While in the ICU
Description: The mean insulin dose during the time that participants were in the ICU is assessed as insulin infusion units per hour.
Time Frame: During the ICU stay (up to 7 days postoperatively)
Population: This analysis includes participants who required CII while in the ICU.
Measure: Mean (Standard Deviation); unit: insulin units/hour
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 11 | 12
insulin units/hour | 2.89 (2.60) | 2.01 (0.98)

7. Secondary Outcome: Mean Insulin Dose Per Day While in the ICU
Description: The mean insulin dose during the time that participants were in the ICU is assessed as insulin units per day.
Time Frame: During the ICU stay (up to 7 days postoperatively)
Population: This analysis includes participants who required CII while in the ICU.
Measure: Mean (Standard Deviation); unit: insulin units/day
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 11 | 12
insulin units/day | 61.15 (66.84) | 33.01 (20.19)

8. Secondary Outcome: Duration of Continuous Insulin Infusion (CII)
Description: The duration of continuous insulin infusion (CII) is assessed in hours.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who required CII while in the ICU.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 11 | 12
hours | 18.90 (5.60) | 16.69 (6.31)

9. Secondary Outcome: Days of Subcutaneous (SC) Insulin After Discontinuation of CII
Description: Subcutaneous (SC) insulin use after continuous insulin infusion (CII) is discontinued is assessed as the number of days that SC insulin was required.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who required CII while in the ICU and subsequent SC after discontinuation of CII.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 6 | 4
days | 2.00 (1.09) | 3.50 (2.08)

10. Secondary Outcome: Amount of SC Insulin Administered
Description: The amount of subcutaneous (SC) insulin administered during the ICU and non-ICU hospital stay, among participants requiring SC insulin after discontinuing CII.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who required CII while in the ICU and subsequent SC after discontinuation of CII.
Measure: Mean (Standard Deviation); unit: units of insulin
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 6 | 4
units of insulin | 8.25 (14.28) | 10.92 (10.44)

11. Secondary Outcome: Number of Participants Experiencing Hyperglycemic Events
Description: Hyperglycemic events are defined as BG > 200 mg/dl, during ICU and non-ICU hospital stay.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
Participants | 1 | 2

12. Secondary Outcome: Number of Participants Experiencing Hypoglycemic Events
Description: Hypoglycemic events are defined as BG <70, < 54, and <40 mg/dl occurring during ICU and non-ICU hospital stay.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
Participants
  BG <70 mg/dL | 0 | 0
  BG <54 mg/dL | 0 | 0
  BG <40 mg/dL | 0 | 0

13. Secondary Outcome: Number of Participants Experiencing Mortality and Complications
Description: The number of participants experiencing a composite of mortality and complications. Complications include sternal wound infection, bacteremia, pneumonia, acute kidney injury, and acute myocardial infarction.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
Participants | 2 | 1

14. Secondary Outcome: Number of Participants Experiencing Gastrointestinal Adverse Events
Description: The number participants who experienced gastrointestinal adverse events of nausea, vomiting, ileus, pancreatitis.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
Participants | 3 | 1

15. Secondary Outcome: ICU Length of Stay
Description: ICU length of stay is assessed as the mean number of days participants in each study arm spent in the ICU.
Time Frame: During the ICU stay (up to 7 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
days | 2.19 (1.45) | 2.76 (1.59)

16. Secondary Outcome: Hospital Length of Stay
Description: Hospital length of stay is assessed as the mean number of days participants in each study arm spent in the hospital.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
days | 7.25 (2.92) | 8.92 (3.72)

17. Secondary Outcome: Number of ICU Readmissions
Description: The number of readmissions to the ICU.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Number; unit: ICU readmissions
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
ICU readmissions | 0 | 0

18. Secondary Outcome: Number of Cerebrovascular Events
Description: The number of cerebrovascular events.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Number; unit: cerebrovascular events
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
cerebrovascular events | 0 | 0

19. Secondary Outcome: Participant Mortality
Description: The number of participant deaths while in the ICU and hospital.
Time Frame: During the hospital stay (up to 12 days postoperatively)
Population: This analysis includes participants who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Dulaglutide | Placebo
Number analyzed (Participants) | 12 | 13
Participants
  ICU deaths | 0 | 0
  Non-ICU hospital deaths | 0 | 0

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected among participants who had elective CABG surgery, beginning at the time of consent and continued through the final assessment occurring 30 days after discharge from the hospital, up to 42 days postoperatively.
Description: Information was collected for the following specific adverse events:sternal wound infection, bacteremia, pneumonia, acute kidney injury, acute myocardial infarction, nausea, vomiting, ileus, and pancreatitis.
Arm/Group | Dulaglutide | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/13
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/13
Other Adverse Events (participants affected / at risk) | 4/12 | 2/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dulaglutide (N=12) | Placebo (N=13)
Hospital readmission due to nausea and vomitting, acute kidney injury, and dehydration (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dulaglutide (N=12) | Placebo (N=13)
Nausea (Gastrointestinal disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-07-30): https://cdn.clinicaltrials.gov/large-docs/25/NCT03743025/Prot_SAP_001.pdf
  • Informed Consent Form (2023-06-21): https://cdn.clinicaltrials.gov/large-docs/25/NCT03743025/ICF_000.pdf